CLINICAL TRIAL: NCT03685578
Title: Embotrap eXtraction & Clot EvaLuation & Lesion Evaluation for NeuroThrombectomy
Brief Title: CERENOVUS Neurothrombectomy Devices Registry
Acronym: EXCELLENT
Status: Completed | Type: Observational
Sponsor: Cerenovus, Part of DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CNV_2017_02; NCT05591183 (obsolete NCT alias)
Record Dates: First submitted 2018-09-07; First posted 2018-09-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Stroke
Keywords: Mechanical thrombectomy; EmboTrap; Embovac; Cereglide 71
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — thrombus / clot
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Mechanical Thrombectomy: EmboTrap® Revascularization Device, CERENOVUS Large Bore Catheter/ EMBOVAC Aspiration Catheter, CEREGLIDE 71 Intermediate Catheter
  Interventions: Device: EmboTrap® Revascularization Device; Device: CERENOVUS Large Bore Catheter/ EMBOVAC Aspiration Catheter; Device: CEREGLIDE 71 Intermediate Catheter

INTERVENTIONS:
Device: EmboTrap® Revascularization Device — EmboTrap® Revascularization Device
Device: CERENOVUS Large Bore Catheter/ EMBOVAC Aspiration Catheter — CERENOVUS Large Bore Catheter/ EMBOVAC Aspiration Catheter
Device: CEREGLIDE 71 Intermediate Catheter — CEREGLIDE 71 Intermediate Catheter

SUMMARY:
A post-market registry evaluating the EmboTrap® Revascularization Device, CERENOVUS Large Bore Catheter/ EMBOVAC™ Aspiration Catheter, and CEREGLIDE 71 Intermediate Catheter in acute ischemic stroke patients with confirmed intracranial vessel occlusion.

DETAILED DESCRIPTION:
The objective of this study are to separately assess the effectiveness of the CERENOVUS neurothrombectomy devices (EmboTrap® Revascularization Device, Large Bore Catheter/EMBOVAC Aspiration Catheter, and CEREGLIDE 71 Intermediate Catheter) in a real-world setting, as well as to explore correlations between patient comorbidities, clot characteristics, revascularization rates, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18
2. The participant or the participant's legally authorized representative has signed and dated an Informed Consent Form. In the event that local regulations allow for alternative approaches of consent, these must be fulfilled as approved by the sponsor and site's ethics committee/regulatory authority (if applicable)
3. Participants experiencing acute ischemic stroke with angiographic confirmation of intracranial vessel occlusion
4. A clinical decision has been made to use a CERENOVUS neurothrombectomy device (EmboTrap® Revascularization Device, Large Bore Catheter/ EMBOVAC Aspiration Catheter, or CEREGLIDE 71 Intermediate Catheter) independently and prior to enrollment in the research study
5. A CERENOVUS neurothrombectomy device is the first attempted primary device/technique for mechanical thrombectomy for the intracranial occlusion in the participant. The following primary devices/techniques are eligible for this study: a) EmboTrap® Revascularization Device alone b) EmboTrap® Revascularization Device + co-aspiration with the Large Bore Catheter/EMBOVAC Aspiration Catheter or CEREGLIDE 71 Intermediate Catheter c) EmboTrap® Revascularization Device + co-aspiration with any other aspiration catheter d) Large Bore Catheter/EMBOVAC Aspiration Catheter alone (that is, direct aspiration with no stent retriever in the first attempted technique) e) CEREGLIDE 71 Intermediate Catheter alone (that is, direct aspiration with no stent retriever in the first attempted technique)

Exclusion Criteria:

1. Currently participating in an investigational (drug, device, etc) clinical trial that may confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible
2. Confirmation of positive pregnancy test according to site specific standard of care (example, test, verbal communication)
3. Use of multiple stent retrievers on the first pass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Ischemic Stroke patients with angiographic confirmation of intracranial vessel occlusion.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Successful Revascularization | 1 day
  Assess cerebral revascularization using the modified Thrombolysis in Cerebral Infarction (mTICI) score at the end of the procedure.

SECONDARY OUTCOMES:
All-Cause Mortality | 90 days
  Summary of all mortality regardless of cause at 90 days post-procedure.
Symptomatic Intracerebral Hemorrhage | 24 hours
  Rate of intracranial hemorrhage as detected by brain imaging (CT/MR) measured 24 hours after intervention
Functional Independence | 90 days
  Modified Rankin Scale (mRS) of ≤ 2
  Modified Rankin Score (Scale from 0-6):
  0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Siddiqui, MD, PhD, Principal Investigator — University at Buffalo; Tommy Andersson, MD, PhD, Principal Investigator — AZ Groeninge/ Karolinska University Hospital; Raul Nogueira, MD, Principal Investigator — UPMC Stroke Institute
Locations (40):
- United States (30):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Banner Desert Medical Center, Mesa, Arizona
  - Barrow Neurological Institute at St. Joseph's Hospital, Phoenix, Arizona
  - Vascular Neurology of Southern California: Dr. M. Asif Taqi, Thousand Oaks, California
  - Memorial Regional Hospital, Hollywood, Florida
  - Baptist Medical Center, Jacksonville, Florida
  - Lyerly Neurosurgery Baptist Health, Jacksonville, Florida
  - University of Miami- Jackson Memorial Hospital, Miami, Florida
  - Advent Health Orlando, Orlando, Florida
  - Emory School of Medicine at Grady Memorial Hospital, Atlanta, Georgia
  - WellStar Health System, Marietta, Georgia
  - Norton Neurology Institute, Elizabethtown, Kentucky
  - Norton Healthcare, Louisville, Kentucky
  - University of Massachusetts, Worcester, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Jacobs Institute/UB Neurosurgery, Inc., Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Mercy Health St Vincent Medical Center, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Geisinger, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - TNVI, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Semmes Murphey Foundation, Memphis, Tennessee
  - University of Texas Houston, Houston, Texas
  - Texas Stroke Institute, Plano, Texas
- Az Groeninge, Kortrijk, Belgium
- Hopital Roger Salengro - CHU Lille, Lille, France
- Germany (4):
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Universitaetsmedizin Mainz, Mainz
  - Radprax MVZ Nordrhein GmbH, Solingen
- Hadassah Medical Center, Jerusalem, Israel
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
- Charing Cross Hospital, London, United Kingdom

REFERENCES:
- [Derived] Nogueira RG, Andersson T, Haussen DC, Yoo AJ, Hanel RA, Zaidat OO, Hacke W, Jovin TG, Fiehler J, De Meyer SF, Brinjikji W, Doyle KM, Kallmes DF, Liebeskind DS, Virmani R, Kokoszka MA, Inoa V, Humphries W, Woodward KB, Jabbour PM, Francois O, Levy EI, Bozorgchami H, Boor S, Cohen JE, Dashti SR, Taqi MA, Budzik RF, Schirmer CM, Hussain MS, Estrade L, De Leacy RA, Puri AS, Chitale RV, Brekenfeld C, Siddiqui AH. EXCELLENT Registry: A Prospective, Multicenter, Global Registry of Endovascular Stroke Treatment With the EMBOTRAP Device. Stroke. 2024 Dec;55(12):2804-2814. doi: 10.1161/STROKEAHA.124.047324. Epub 2024 Nov 19. PMID 39559856
- [Derived] Bilgin C, Dai D, Johnson C, Mereuta OM, Kallmes DF, Brinjikji W, Kadirvel R. Quality assessment of histopathological stainings on prolonged formalin fixed thrombus tissues retrieved by mechanical thrombectomy. Front Neurol. 2023 Dec 13;14:1223947. doi: 10.3389/fneur.2023.1223947. eCollection 2023. PMID 38152640
- [Derived] Siddiqui AH, Waqas M, Brinjikji W, De Meyer SF, Doyle K, Fiehler J, Hacke W, Hanel RA, Jovin TG, Liebeskind DS, Yoo AJ, Zaidat OO, Andersson T, Nogueira RG. Embotrap Extraction & Clot Evaluation & Lesion Evaluation for NeuroThrombectomy (EXCELLENT) Registry design and methods. J Neurointerv Surg. 2022 Aug;14(8):783-787. doi: 10.1136/neurintsurg-2021-017671. Epub 2021 Oct 13. PMID 34645704